CLINICAL TRIAL: NCT02926781
Title: A Comparative Study to Evaluate Bone Height Gain Following Transcrestal Sinus Floor Elevation Using Specially Designed Drills Versus the Conventional Osteotome Technique: a Randomized Controlled Clinical Trial.
Brief Title: A Comparative Study to Evaluate Bone Height Gain Following Transcrestal Sinus Floor Elevation Using Specially Designed Drills Versus the Conventional Osteotome Technique.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Ashour, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Omar Ashour
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Compromised Vertical Bone Height in the Maxillary Posterior Region

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- osteotome technique (Experimental): transcrestal sinus floor elevation using osteotomes
  Interventions: Device: Dask Advanced Sinus kit
- drills (Active Comparator): transcrestal sinus floor elevation using drills
  Interventions: Device: Dask Advanced Sinus kit

INTERVENTIONS:
Device: Dask Advanced Sinus kit — a kit of specially designed drills for closed sinus lift

SUMMARY:
Radiographic evaluation of the amount of bone height gain and clinical evaluation of the possibility of developing complications after transcrestal sinus floor elevation using drills and the conventional osteotome technique.

DETAILED DESCRIPTION:
Short implants (< 10 mm) are one of the options used to overcome low vertical bone height in the maxilla. However, short implants have faced many challenges as smaller implant surface; therefore less bone-to-implant contact after osseointegration with force distribution on a reduced surface after loading. This leads to more crestal bone resorption with more threads exposure decreasing the long term implant success Another treatment option is placing implants in specific anatomical areas, such as the pterygoid region or the zygoma .Many complications are reported as postoperative sinusitis, temporary paresthesia, epistaxis, facial, periorbital hematoma, orbital penetration and prosthetic difficulties due to the implants palatal emergence.

Vertical augmentation with bone grafts is another treatment option. However, it has many drawbacks as the unpredictable graft resorption, low bone to implant contact, higher possibility of wound dehiscence, as well as compromised implant position leading to undesirable prosthetic restorations.

To overcome the problems of the previously mentioned procedures, elevation of the sinus membrane techniques were proposed, it can be performed either through a lateral window , or via a crestal access depending on the remaining bone height (RBH). If the RBH is around 6-9 mm, the crestal approach is indicated. If the RBH is less than 5 mm, a lateral approach should be performed.

For the crestal approach, it could be performed by the conventional osteotome technique. However, it is a visually restrictive technique which may lead to sinus perforation as well as it can cause some complications as headache and paroxysmal positional vertigo (Saker e Ogle, 2005; Peñarrocha-Diago et al., 2008).

To overcome the disadvantages of the conventional osteotome technique, various kits have been developed for transcrestal sinus floor elevations using specially designed drills.

ELIGIBILITY:
Inclusion criteria

Patients having at least one missing upper posterior tooth.

Residual bone height beneath maxillary sinus from 5-8 mm .

A minimum of 6 mm residual bone width.

The recipient site of the implant should be free from any pathological condition.

No diagnosed bone disease or medication known to affect bone metabolism.

Patients who are cooperative, motivated and hygiene conscious.

Patients having proper inter-occlusal space.

Exclusion criteria

Systemic conditions/disease that contraindicated surgery.

Radiation therapy in the head and neck region or chemotherapy during the 12 months prior to surgery.

Patients who have any habits that might jeopardize the osseointegration process, such as current smokers.

Patients with parafunctional habits that produce overload on implant, such as bruxism and clenching.

Patients that have any pathology in the maxillary sinuses.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
bone height gain | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Omar A Ashour, Bachelor, Principal Investigator — Cairo University